CLINICAL TRIAL: NCT05684419
Title: Observation of the Fate and Quality of Medical Follow-up of Children Born Preterm to Homeless Mothers.
Brief Title: Preterm Infants Born to Homeless Mothers.
Acronym: PREMA-NEUF
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0522
Record Dates: First submitted 2022-12-16; First posted 2023-01-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Prematurity; Extreme
Keywords: Premature; Homeless; Extreme prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Fate and quality of medical follow-up of children born very premature (≤33SA) to homeless mothers — Evaluation of the fate and quality of medical follow-up of children born very premature (≤33SA) to homeless mothers.

SUMMARY:
In recent years, the number of homeless patients who are accommodated by the SAMU social has increased. These patients are in a situation of financial, but also often social and psychological precariousness. The literature already shows us that precariousness and homelessness are a risk factor for prematurity, but also for the patients themselves, a risk of more frequent recourse to emergency services and of late consultation for advanced pathologies.

The objective of this study is to evaluate the fate and quality of medical follow-up of children born very premature (≤33SA) to homeless mothers.

DETAILED DESCRIPTION:
The hospital of Pontoise is the largest maternity hospital in the department (Val d'Oise, 95) with 4449 births in 2021. It has a type 3 neonatal intensive care unit where approximately 150 premature babies under 32 weeks of age are hospitalized each year, including 80 premature babies under 28 weeks of age. These children require a specific and prolonged follow-up after hospitalization, including medical consultations to evaluate their neurodevelopmental development, but also the prevention of RSV infection (Respiratory Syncitial Virus).

In recent years, the number of homeless patients who are accomodated by the SAMU social has increased. These patients are in a precarious financial, but also often social and psychological situation. The literature already shows us that precariousness and homelessness are a risk factor for prematurity, but also for the patients themselves, a risk of more frequent recourse to emergency services and late consultation with advanced pathologies.

The aim of this study is to evaluate the fate and quality of medical follow-up of children born very premature (≤33SA) to homeless mothers, by answering the following questions:

* What about the follow-up of their very premature child?
* How does the department organize itself to ensure optimal follow-up for these patients?

ELIGIBILITY:
Inclusion Criteria :

All infants born at or below 33SA:

* Born between January 2019 and December 2021
* At the René Dubos Hospital in Pontoise
* Whose mother did not have a fixed address at the time of discharge.

NB: Mothers who do not read French well will have the study explained to them by the doctor who follows their child during a consultation, or by telephone.

Exclusion Criteria :

- Opposition of the mothers

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants born at or below 33SA:
  * Born between January 2019 and December 2021
  * At the René Dubos Hospital in Pontoise
  * Whose mother did not have a fixed address at the time of discharge.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Assessment of the rate of infants born to homeless mothers at or below 33 SA and lost to follow-up for extreme prematurity | At 12 month
  Measurement of the number of children lost to follow-up at 12 months who missed their last follow-up appointment(s) organized in the context of prematurity, with no reason given or new schedule planned

SECONDARY OUTCOMES:
Assessment of the compliance of homeless mothers with medical prescriptions and the respect of the instructions given for the course of care (treatments, physiotherapy, appointment scheduling, etc.) | At 12 month
  Measurement of the compliance rate of homeless mothers with medical prescriptions (treatments, physical therapy, appointment scheduling, etc.) at 12 months
Assessment of vaccination rates in infants born at or below 33 days' gestation to homeless mothers | At 12 month
  Measure of the number of children with full immunization among children born at 33 SA or less to homeless mothers at 12 months
Assessment of the organized follow-up in the city of infants born at a term less than or equal to 33 days of age, of homeless mothers (between the PMI and the attending physicians) | At 6 month
  Description of the type of organized follow-up in town of infants born at a term less than or equal to 33 days of age, of homeless mothers (between the PMI and the attending physicians, spacing of appointments), evaluated at 6 months
Assessment of the rate of re-hospitalization and consultation in the emergency room of the René Dubos Hospital for infants born at a term less than or equal to 33 days of age, of homeless mothers | At 12 month
  Measurement of the number of re-hospitalizations and emergency room visits at the René-Dubos Hospital for infants born at a term of less than or equal to 33 weeks of age, to homeless mothers, evaluated at 12 months
Assessment of breastfeeding duration at 6 months in infants born at or below 33 days' gestation to homeless mothers | At 6 month
  Measurement of breastfeeding duration in weeks, assessed at 6 months, in infants born at or below 33 SA to homeless mothers
Assessment of the type of feeding on the duration of follow-up in infants born at a term less than or equal to 33 SA, of homeless mothers | At 12 month
  Description of the type of feeding (breastfeeding, industrial milk, diversification) in infants born at a term less than or equal to 33 SA, of homeless mothers
Assessment of staturo-weight growth during follow-up in infants born at or below 33 SA born to homeless mothers | At 12 month
  Analysis of the staturo-weight growth curve (weight and Z score) in infants born at a term of less than or equal to 33 SA, to homeless mothers

CONTACTS AND LOCATIONS:
Overall Officials: Dr Suzanne BORRHOMEE, Principal Investigator — Hôpital NOVO
Locations (1):
- Resuscitation and neonatal medicine department - Centre Hospitalier René Dubos, Pontoise, France

IPD SHARING:
Plan to Share IPD: No